CLINICAL TRIAL: NCT05702827
Title: Use of a Dual-agent Local Analgesic (Bupivacaine-meloxicam) for Abdominal Incisions in Patients Undergoing Retropubic Mid-urethral Sling Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-102
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Stress Urinary Incontinence; Surgical Incision; Pain Vulva
MeSH Terms: conditions — Urinary Incontinence, Stress; Surgical Wound; Vulvodynia | interventions — bupivacaine-meloxicam drug combination

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- bupivacaine-meloxicam (Experimental): All patients will receive a total of 20 cc lidocaine with epinephrine injection intra-operatively along the trocar path via the suprapubic incisions, as is standard practice to help with hydrodissection for the procedure. 3-4 cc of bupivacaine-meloxicam will be infiltrated into each suprapubic abdominal incision in the study group
  Interventions: Drug: Bupivacaine-Meloxicam
- Standard of Care (No Intervention): All patients will receive a total of 20 cc lidocaine with epinephrine injection intra-operatively along the trocar path via the suprapubic incisions, as is standard practice to help with hydrodissection for the procedure.

INTERVENTIONS:
Drug: Bupivacaine-Meloxicam — All patients will receive standard of care but the study arm will also receive Bupivacaine-Meloxicam in addition.
  Arms: bupivacaine-meloxicam

SUMMARY:
This study will compare the use of a dual-agent local analgesic (bupivacaine-meloxicam) for abdominal incisions in patients undergoing retropubic mid-urethral sling surgery to see if narcotic usage and pain are impacted.

ELIGIBILITY:
Inclusion Criteria:

* undergoing retropubic mid-urethral sling surgery (with concomitant anterior repair or urethrocele repair)
* English as first language

Exclusion Criteria:

* patients undergoing concomitant posterior repair, vaginal vault suspension, or any other intra-peritoneal surgeries including hysterectomy
* NSAID use within 7 days of surgery
* steroid use within 10 days
* daily opioid use in the last 3 months
* long acting opioids within 3 days
* any opioids within 24h
* patients unable to consent for themselves
* patients allergic to meloxicam or bupivacaine
* pregnant or lactating patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
To determine if use of bupivacaine-meloxicam reduces post-operative narcotic use over the first 3 days following surgery | 72 hours post surgery
  Pain medication diary

SECONDARY OUTCOMES:
Compare average pain on each day post operatively | 72 hours post surgery
  11-point Numeric Rating Scale (NRS) for tracking pain using an illustrated figure to localize the pain, a 5-point Likert scale for satisfaction with pain control a Quality of Recovery (QoR-15) questionnaire filled out before surgery and on post-operative days 1 and 3
Compare worst pain on each day post operatively | 72 hours post surgery
  11-point Numeric Rating Scale (NRS) for tracking pain using an illustrated figure to localize the pain, a 5-point Likert scale for satisfaction with pain control a Quality of Recovery (QoR-15) questionnaire filled out before surgery and on post-operative days 1 and 3
Compare satisfaction with pain control post operatively | 72 hours post surgery
  11-point Numeric Rating Scale (NRS) for tracking pain using an illustrated figure to localize the pain, a 5-point Likert scale for satisfaction with pain control a Quality of Recovery (QoR-15) questionnaire filled out before surgery and on post-operative days 1 and 3

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cincinnati Urogynecology Associates, Cincinnati, Ohio
  - Trihealth (Good Samaritan Hospital, Bethesda North Hospital), Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No